CLINICAL TRIAL: NCT00603629
Title: A Pilot Study Determining Mechanisms of Acute Asthma Exacerbations Through Detailed Molecular Analysis of Airway Secretions and Tissues
Brief Title: Mechanisms of Acute Asthma Exacerbations Through Molecular Analysis of Airway Secretions and Tissues
Acronym: MAST-X
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, John V. Fahy, Professor in Residence, University of California, San Francisco
Other Study IDs: H6788-31516-01
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Asthma
Keywords: Acute Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, DNA, RNA, sputum, nasopharyngeal swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- I: People with acute asthma in the Emergency department or inpatient settings

SUMMARY:
The purpose of this study is to investigate mechanisms which cause acute asthma exacerbations by examining blood and airway secretions during an acute onset (sputum or tracheal aspirates). This pilot study is intended to uncover new mechanisms of asthma exacerbation and to generate hypotheses for future study. By collaborating with Genentech, we (scientists at UCSF) plan to incorporate the latest scientific findings into our work to discover and develop new treatments for asthma.

DETAILED DESCRIPTION:
Asthma is a common airway disease with persistent unmet needs in terms of treatment. Although many asthmatics enjoy good control of their disease by using regularly scheduled corticosteroid treatment, a significant minority do not achieve optimal control with steroids and suffer asthma exacerbations which can be severe and even fatal. Asthma pathophysiology is complex and involves multiple cell types and multiple signaling mechanisms. One approach to this complexity has been to study responses of isolated airway cells to experimental conditions which model asthmatic inflammation; another has been genetic manipulations of candidate mediators of asthma in inbred mice. These studies have yielded important insights about possible mechanisms of asthma in humans, but the relevance of these mechanisms to human disease has not always been proven, and it is possible that unsuspected mechanisms have not yet been revealed by these approaches.

In the current study, we propose to collect samples of airway secretions and blood from asthmatic subjects when their asthma is uncontrolled and they are being treated in the hospital or emergency room. Our goal will be to identify abnormal gene expression profiles and protein concentration abnormalities in these biological fluids. We will then study them again 6-10 weeks later when their asthma is controlled. This study design will allow us to compare airway and blood biomarkers of asthma exacerbation during acute asthma and recovery. "

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 - 70 years
2. Medical history of asthma
3. Currently experiencing an acute exacerbation of asthma
4. Ability to provide informed consent or have a surrogate provide consent.
5. Ability to provide sputum.

Exclusion Criteria:

1. Cigarette smoking: Subjects must be non-smokers. Non-smokers are defined as subjects who have never smoked or who have not smoked for 1 year and have a total pack-year smoking history < 10 packs.
2. Pregnant women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with acute asthma who seek treatment in the Emergency Department or who require admission to the hospital for their asthma
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

SECONDARY OUTCOMES:
gene expression in acute airway secretions and tissues | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: John V Fahy, M.D., M.Sc., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

REFERENCES:
- See also: UCSF Airway Clinical Research Center website — http://airway.ucsf.edu